CLINICAL TRIAL: NCT06417983
Title: Use of Topical Essential Oil Compound to Treat Toe Nail Onychomycosis
Brief Title: Topical Application of Essential Oils to Treat Onchomycosis
Acronym: NailFungus
Status: Not yet recruiting | Type: Observational
Sponsor: Medical Life Care Planners, LLC (Other)
Responsible Party: Principal Investigator, Gregory L Smith, MD, MPH, Principal Investigaor, Medical Life Care Planners, LLC
Other Study IDs: Onychomycosis Topical
Record Dates: First submitted 2024-04-23; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Onychomycosis of Toenail; Fungal Infection; Toenail Infection
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with documented onychomycosis of one or more toe nails will be treated with a daily application of a topical lacquer containing several essential oils.

DETAILED DESCRIPTION:
The topical lacquer contains the following components:

Active ingredients:

Hydroxypropyl Chitosan OLEOZON(r) - natural, ozonized sunflower oil. Vitamin E Tea Tree Oil Cannabidiol

Vehicle:

Nanoparticle medium chain triglyceride oil

ELIGIBILITY:
Inclusion Criteria:

Clinician observation consistent with probable onychomycosis of one or more toenails.

Positive polymerase chain reaction (PCR) for fungal infection or Positive Periodic Acid Schiff, Biopsy, KOH or Culture for fungal infection -

Exclusion Criteria:

Unwlling to discontinue current anti-fungal medication, oral or topical

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting to a community podiatry clinic who upon examination are noted to have podiatrist diagnosed onychomycosis of one or more toenails. Not currently using topical or oral anti-fungal treatment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Thickness of the Hyponychium Fungal Infection | 12 weeks
  Objective change in the thickness of the hyponychium of the most infected nailplate. The hyponycium will be measured with a micometer thickness guage in micrometer gradations at baseline, 2,5,9 and 12 weeks.
Subject Perceived Improvement in overall toenail infection | 12 weeks
  Subject's personal perception of improvement of all infected toenails using the OnyCOE-t questionnaire for patient reported outcomes for toenail onychomycosis at baseline, 2,5 ,9 and 12 weeks of treatment.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months
Access Criteria: Researcher with clear need to know
URL: http://nex-therapeutics.com

REFERENCES:
- [Background] Flores FC, Beck RC, da Silva Cde B. Essential Oils for Treatment for Onychomycosis: A Mini-Review. Mycopathologia. 2016 Feb;181(1-2):9-15. doi: 10.1007/s11046-015-9957-3. Epub 2015 Oct 19. PMID 26481920
- [Background] Halteh P, Scher RK, Lipner SR. Over-the-counter and natural remedies for onychomycosis: do they really work? Cutis. 2016 Nov;98(5):E16-E25. PMID 28040821
- [Background] Wang Y, Lipner SR. Retrospective analysis of adverse events with topical onychomycosis medications reported to the United States Food and Drug Administration. Arch Dermatol Res. 2020 Oct;312(8):581-586. doi: 10.1007/s00403-020-02044-7. Epub 2020 Feb 19. PMID 32076805
- [Background] Abd Rashed A, Rathi DG, Ahmad Nasir NAH, Abd Rahman AZ. Antifungal Properties of Essential Oils and Their Compounds for Application in Skin Fungal Infections: Conventional and Nonconventional Approaches. Molecules. 2021 Feb 19;26(4):1093. doi: 10.3390/molecules26041093. PMID 33669627
- [Background] Ghannoum MA, Long L, Isham N, Bulgheroni A, Setaro M, Caserini M, Palmieri R, Mailland F. Ability of hydroxypropyl chitosan nail lacquer to protect against dermatophyte nail infection. Antimicrob Agents Chemother. 2015 Apr;59(4):1844-8. doi: 10.1128/AAC.04842-14. Epub 2014 Dec 29. PMID 25547349
- [Background] Feldman M, Sionov RV, Mechoulam R, Steinberg D. Anti-Biofilm Activity of Cannabidiol against Candida albicans. Microorganisms. 2021 Feb 20;9(2):441. doi: 10.3390/microorganisms9020441. PMID 33672633
- [Background] Tong MM, Altman PM, Barnetson RS. Tea tree oil in the treatment of tinea pedis. Australas J Dermatol. 1992;33(3):145-9. doi: 10.1111/j.1440-0960.1992.tb00103.x. PMID 1303075